CLINICAL TRIAL: NCT05483101
Title: Accompagnement de la Grossesse et de la Naissance en filière Physiologique Par Rapport en filière Conventionnelle : Effet Sur la Voie d'Accouchement et la santé périnatale
Brief Title: Personalized Support Care in Alternative Midwifery Birth Units Versus Traditional Units in France : Effects on Perinatal Health and Outcomes
Acronym: PhysioCare
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC20_8988_PhysioCare
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Compare 2 Models of Midwifery Care in Maternity Care
Keywords: Midwife-led care; midwifery birth units; physiologic birth; continuity of patient care; humanized care; quality of health care; safety

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- alternative units: In alternative birth units : personalized follow-up with a midwife from the beginning of pregnancy, birth and parenthood preparation classes and delivery (birth room).
  Interventions: Other: Alternative birth units
- conventional units: In standard maternity care, most full time midwives are rostered to work. They follow women during their pregnancy but not through labour. All low-risk pregnant women benefit from 5 prenatal consultations with a general practitioner, a midwife or an obstetrician, then 2 consultations with a midwife in maternity hospital of delivery. Couples have got the option to elaborate a birth project if desired

INTERVENTIONS:
Other: Alternative birth units — Midwife-led alternative birth units are a new model of care in France in which the midwife is the primary health care professional caring for low-risk pregnant women, as opposed to those cared for by an obstetrician-led medical team. Accordingly, alternative birth units also provide a space within which midwives can practice to their fullest potential with more professional autonomy than in a traditional obstetric setting. These birth units emphasizes care that promotes normal physiologic pregnancy and labor and supports the natural ability of women to experience birth with minimum or no routine intervention.
  Alternative birth units named "Filière physiologique (FP) co-exist in the same building on the same site as a hospital or host obstetric unit. In the event a laboring women needs comprehensive emergency obstetric care, she can be transferred immediatly in a conventionnal birth room.
  Groups: alternative units

SUMMARY:
Most pregnancies and deliveries in France occur without complication. According to the 2016 Perinatal Survey, 2/3 of births are carried out by spontaneous vaginal delivery with midwife support in most cases. Although the impact of lack of care is now well recognized, literature reveals that overmedicalization of pregnancy and birth follow-up is not associated with better health outcomes for women and children. Rather, it may have a deleterious impact, in addition to unnecessary health care costs. Recent national and international guidelines in the management of normal childbirth support the facilitation of physiologic labor and the minimization of non-medically justified interventions, particularly for women at low obstetric risk.

Providing specific places to support low-rick pregnant women is an opportunity to preserve physiology.

In France, 4 innovative care units called Filières Physiologiques (FP), have been developed on an experimental model within hospital structures in recent years. The FPs, unlike freestanding midwifery units, allow a non-medicalized birth within a maternity hospital, with immediate care of the pregnant women and/or their child in case of vital emergency. A personalized follow-up with a midwife from the beginning of the pregnancy, birth and parenthood preparation classes and delivery is proposed to couples wishing to.

Existing studies in France and abroad show that support outside the conventional care network does not increase perinatal morbidity and improves the experience of childbirth, with a positive influence on the establishment of the mother-child bond and the psychological state of the parents in postpartum. In addition, several studies conducted abroad suggest that follow-up by a midwife could reduce the costs of perinatal care for the health system. However, these studies were conducted abroad, with different structures of follow-up in FP.

A care approach, as proposed in the FPs, with physiological accompaniment of childbirth by a midwife who is available and listens to the couple (the "one-to-one" principle with individual support for the woman) would improve the experience of couples, reduce the stress, fear and pain of labor, and diminish the feeling of insecurity. Other studies suggest that psychosomatic support during pregnancy could reduce the risk of postpartum depression, which is a public health issue.

This study suggest that FP care for women at low obstetrical risk, as compared with conventionnal birth care unit, would promote spontaneous vaginal birth without instrumental extraction. Another hypothesis is that this management would improve salutogenesis indicators, the birth experience of couples, the establishment of the mother-child bond, and the psychological state of parents in the postpartum period. FP care could also be more efficient than conventionnal birth care unit from the community's perspective.

DETAILED DESCRIPTION:
This study consists in a prospective multicenter cohort, exposed/unexposed, recruiting 567 low-risk pregnant women in 3 French maternity hospitals from septembre 2022, between 34 and 39 weeks of amenorrhea, matched by center and parity (189 in alternative units and 378 in conventional units). Data will be collected from medical record and questionnaires completed by women and partners at inclusion, 2 days, 3 and 6 weeks postpartum (Mother-to-Infant Bonding Scale; Maternal Childbirth Experience Assessment Questionnaire; First-Time Father Questionnaire; Peritraumatic Distress Inventory; Impact of Event Scale-Revised; Edinburgh Postnatal Depression Scale). Semi-structured interviews to assess women's, partners' and professionals' perceptions of care will be conducted on a sample of couples and midwives. Costs included all costs to the health system for the whole pregnancy up to 6 weeks postpartum, and outcomes will be quality-adjusted life years (QALY) gained. Multivariate intention-to-treat statistical analyses (linear/logistic regression with propensity score, IPTW) will be performed.

Benefits to families through increased knowledge of midwifery care's impact on birth process and parents' birth experience.

This could allow for expansion of alternative birth units in other health care settings.

ELIGIBILITY:
Inclusion Criteria:

* Low-risk pregnancy according to the HAS clinical practice recommendations (2016): follow-up classified A (without particularity) provided indifferently by a FS or a physician; eligibility if follow-up classified A1 or A2 after advice from an ob-gyn and/or another specialist.
* Gestational age between 34 and 39 weeks of amenorrhea
* Single pregnancy
* Maternal age ≥ 18 et < 40 years old
* Patient who planned to give birth in a maternity hospital involved in the study.
* Having been informed about the protocol and not having expressed opposition to participate in the PhysioCare study.

Non-inclusion criteria:

* Psychiatric history or depression with medication
* Anonymous childbirth
* History of caesarean section
* Undeclared pregnancy, not or poorly followed up (no blood/urinary check-ups carried out during pregnancy and/or no monthly follow-up with medical consultation)
* Couples unable to speak French
* Non-affiliation of patient to a social security scheme
* Adult persons subject to legal protection ; persons deprived of their liberty

Exclusion Criteria:

* Fetal death or medical termination of pregnancy after inclusion
* Death of the child at birth
* Premature birth < 37 weeks of age

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who planned to give birth in a maternity hospital involved in the study, with a low risk pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Mode of delivery according to care of pregnant women in alternative midwifery birth units versus traditional birth units | up to 5 weeks
  Rate of spontaneous vaginal delivery versus instrumental vaginal delivery and cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Ronan GARLANTEZEC, Principal Investigator — Rennes University Hospital
Locations (3):
- France (3):
  - Centre Hospitalier Simone Veil, Eaubonne
  - Clinique Mutualiste La Sagesse, Rennes
  - Rennes University Hospital, Rennes

IPD SHARING:
Plan to Share IPD: No